CLINICAL TRIAL: NCT02310581
Title: A Phase 3, Randomized, Double-Blind, Multiple-Dose, Parallel-Group, Placebo-Controlled Study of Buprenorphine Sublingual Spray for the Treatment of Moderate to Severe Pain
Brief Title: Buprenorphine Sublingual Spray for the Treatment of Moderate to Severe Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS-14-026
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-06

CONDITIONS: Post-operative Pain
Keywords: Bunionectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Buprenorphine 0.5 mg TID (Experimental): Participants received buprenorphine 0.5 mg sublingual spray three times daily (TID) and placebo-matching buprenorphine sublingual spray once daily (QD) for two days.
  Interventions: Drug: Buprenorphine Sublingual Spray; Drug: Placebo
- Buprenorphine 1.0 mg BID (Experimental): Participants received buprenorphine 1.0 mg sublingual spray twice daily (BID) and placebo-matching buprenorphine sublingual spray BID for two days.
  Interventions: Drug: Buprenorphine Sublingual Spray; Drug: Placebo
- Buprenorphine 1.0 mg TID (Experimental): Participants received buprenorphine 1.0 mg sublingual spray TID and placebo-matching buprenorphine sublingual spray QD for two days.
  Interventions: Drug: Buprenorphine Sublingual Spray; Drug: Placebo
- Placebo (Placebo Comparator): Participants received placebo-matching buprenorphine sublingual spray four times daily for two days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine Sublingual Spray — Buprenorphine sublingual spray delivered via single 100 μL spray
  Arms: Buprenorphine 0.5 mg TID; Buprenorphine 1.0 mg BID; Buprenorphine 1.0 mg TID
Drug: Placebo — Placebo-matching buprenorphine sublingual spray delivered via single 100 μL spray

SUMMARY:
This is a phase 3, multicenter, randomized, double-blind, multiple-dose, parallel-group, placebo-controlled study to evaluate the safety and efficacy of up to 3 dosing regimens of Buprenorphine Sublingual (under the tongue) Spray and/or matching placebo in participants with moderate to severe postoperative pain after bunionectomy. The study will comprise 4 periods: the Screening Period, the Surgical Period, the Treatment Period, and the Follow-up Period.

Participants will be admitted to the study site on the morning of the scheduled surgery, will remain at the study site until postoperative Day 3 (a total of 3 nights at the study site), and will return for the Follow-up Visit 5 to 9 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Is able to speak and understand the language in which the study is being conducted, is able to understand the procedures and study requirements and has voluntarily signed and dated an informed consent form approved by the Institutional Review Board before the conduct of any study procedure
* Is willing and able to comply with study requirements (including diet, alcohol, and smoking restrictions), complete the pain evaluations, remain at the study site for three days, and return for follow up between 7 and 9 days after surgery.

Exclusion Criteria:

* History or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2015-03-19 (Actual); Study Completion 2015-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni DeCastro, Study Director — INSYS Therapeutics Inc
Locations (3):
- United States (3):
  - Phoenix, Arizona
  - Pasadena, Maryland
  - Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine 0.5 mg TID: Participants received buprenorphine 0.5 mg sublingual (under the tongue) spray three times daily (TID) and placebo-matching buprenorphine sublingual spray once daily (QD) for two days.
Period: Overall Study
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Started | 9 | 11 | 10 | 10
Completed | 6 | 9 | 9 | 9
Not Completed | 3 | 2 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo | Total
Number analyzed (Participants) | 9 | 11 | 10 | 10 | 40
Age, Continuous [Mean (Full Range); unit: years] | 48.0 [31.0 to 65.0] | 43.5 [26.0 to 65.0] | 40.8 [28.0 to 61.0] | 40.5 [19.0 to 61.0] | 43.2 [19.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 7 | 9 | 32
  Male | 2 | 2 | 3 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Summed Pain Intensity Difference (SPID) Over 0 to 48 Hours After Time 0 (NRS SPID-48)
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug) and at multiple time points up to 48 hours after Time 0 (administration of first dose of study drug). Pain intensity difference is calculated by subtracting the pain intensity at each time point from the pain intensity at Time 0. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [maximum (max)=10 at each time point] and negative numbers indicate an increase in pain [minimum (min)=-10 at each time point]. The overall min and max are -10 and 10 times the number of hours specified; SPID-48 range is -480 to 480. The NRS SPID-48 was analyzed using an analysis of covariance (ANCOVA) model, which included treatment and site as main effects and Baseline pain intensity as the covariate.
Time Frame: Baseline and 0 to 48 hours after Time 0
Population: All randomized participants from the Intent-to-Treat (ITT) Population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 10
units on a scale | 169.621 (29.9942) | 150.964 (27.5418) | 129.133 (29.3429) | 64.648 (29.0597)
Statistical Analysis 1: Comparison: Buprenorphine 0.5 mg TID vs Placebo; Test type: Other; p = 0.012, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 104.973, 95% CI 2-sided [25.13 to 184.81], Standard Error of Mean 39.2433
Statistical Analysis 2: Comparison: Buprenorphine 1.0 mg BID vs Placebo; Test type: Other; p = 0.028, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 86.316, 95% CI 2-sided [9.94 to 162.69], Standard Error of Mean 37.5385
Statistical Analysis 3: Comparison: Buprenorphine 1.0 mg TID vs Placebo; Test type: Other; p = 0.110, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 64.485, 95% CI 2-sided [-15.36 to 144.33], Standard Error of Mean 39.2459

2. Secondary Outcome: NRS Mean Pain Intensity Difference (PID) at 4, 8, 24 and 48 Hours After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug administration) and at multiple time points up to 48 hours after Time 0 (time of administration of the first dose of study drug). NRS PID is defined as the difference in pain at each scheduled timepoint relative to Baseline (PID=pain intensity at baseline - pain intensity at time point). A higher value of NRS PID score indicates a higher decrease in pain from Baseline.
Time Frame: Baseline and 4, 8, 24 and 48 hours after Time 0
Population: All randomized participants from the ITT Population with data available at each timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 10
units on a scale
  4 Hours: number analyzed (Participants) | 9 | 11 | 10 | 9
  4 Hours | 4.7 (1.73) | 3.4 (3.01) | 3.8 (2.94) | 1.6 (1.33)
  8 Hours: number analyzed (Participants) | 8 | 11 | 10 | 9
  8 Hours | 3.4 (1.41) | 4.0 (2.97) | 3.9 (2.28) | 1.2 (1.99)
  24 Hours: number analyzed (Participants) | 6 | 9 | 9 | 9
  24 Hours | 5.5 (1.76) | 3.0 (3.16) | 3.4 (1.81) | 2.6 (1.94)
  48 Hours: number analyzed (Participants) | 6 | 9 | 9 | 9
  48 Hours | 6.3 (1.03) | 4.2 (2.39) | 4.1 (2.80) | 3.2 (2.64)

3. Secondary Outcome: NRS Mean Pain Intensity Score at 4, 8, 24 and 48 Hours After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug administration) and at multiple time points up to 48 hours after Time 0 (time of administration of the first dose of study drug). A lower value indicates improvement in pain.
Time Frame: 4, 8, 24 and 48 hours after Time 0
Population: All randomized participants from the ITT Population with data available at each timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 10
units on a scale
  4 Hours: number analyzed (Participants) | 9 | 11 | 10 | 9
  4 Hours | 2.2 (2.49) | 2.9 (3.08) | 4.0 (2.87) | 4.9 (3.14)
  8 Hours: number analyzed (Participants) | 8 | 11 | 10 | 9
  8 Hours | 3.5 (2.14) | 2.3 (3.00) | 3.9 (2.42) | 5.2 (2.64)
  24 Hours: number analyzed (Participants) | 6 | 9 | 9 | 9
  24 Hours | 1.8 (1.47) | 3.3 (2.55) | 4.6 (2.07) | 3.9 (2.80)
  48 Hours: number analyzed (Participants) | 6 | 9 | 9 | 9
  48 Hours | 1.0 (0.89) | 2.1 (1.76) | 3.9 (2.42) | 3.2 (2.11)

4. Secondary Outcome: NRS SPID Over 0 to 4 Hours After Time 0 (NRS SPID-4)
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug) and at multiple time points up to 4 hours after Time 0 (administration of first dose of study drug). Pain intensity difference is calculated by subtracting the pain intensity at each time point from the pain intensity at Time 0. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [maximum (max)=10 at each time point] and negative numbers indicate an increase in pain [minimum (min)=-10 at each time point]. The overall min and max are -10 and 10 times the number of hours specified; SPID-4 range is -40 to 40. The NRS SPID-4 was analyzed using an analysis of covariance (ANCOVA) model, which included treatment and site as main effects and Baseline pain intensity as the covariate.
Time Frame: Baseline and 0 to 4 hours after Time 0
Population: ITT Population included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 10
units on a scale | 11.430 (3.6221) | 5.088 (3.3259) | 7.095 (3.5434) | -2.968 (3.5092)
Statistical Analysis 1: Comparison: Buprenorphine 0.5 mg TID vs Placebo; Test type: Other; p = 0.005, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 14.398, 95% CI 2-sided [4.76 to 24.04], Standard Error of Mean 4.7390
Statistical Analysis 2: Comparison: Buprenorphine 1.0 mg BID vs Placebo; Test type: Other; p = 0.085, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 8.056, 95% CI 2-sided [-1.17 to 17.28], Standard Error of Mean 4.5331
Statistical Analysis 3: Comparison: Buprenorphine 1.0 mg TID vs Placebo; Test type: Other; p = 0.041, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 10.063, 95% CI 2-sided [0.42 to 19.70], Standard Error of Mean 4.7393

5. Secondary Outcome: NRS SPID Over 0 to 8 Hours After Time 0 (NRS SPID-8)
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug) and at multiple time points up to 8 hours after Time 0 (administration of first dose of study drug). Pain intensity difference is calculated by subtracting the pain intensity at each time point from the pain intensity at Time 0. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [maximum (max)=10 at each time point] and negative numbers indicate an increase in pain [minimum (min)=-10 at each time point]. The overall min and max are -10 and 10 times the number of hours specified; SPID-8 range is -80 to 80. The NRS SPID-8 was analyzed using an analysis of covariance (ANCOVA) model, which included treatment and site as main effects and Baseline pain intensity as the covariate.
Time Frame: Baseline and 0 to 8 hours after Time 0
Population: ITT Population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 10
units on a scale | 24.283 (6.2667) | 19.223 (5.7543) | 19.761 (6.1306) | -2.382 (6.0715)
Statistical Analysis 1: Comparison: Buprenorphine 0.5 mg TID vs Placebo; Test type: Other; p = 0003, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 26.665, 95% CI 2-sided [9.98 to 43.35], Standard Error of Mean 8.1991
Statistical Analysis 2: Comparison: Buprenorphine 1.0 mg BID vs Placebo; Test type: Other; p = 0.009, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 21.605, 95% CI 2-sided [5.65 to 37.56], Standard Error of Mean 7.8429
Statistical Analysis 3: Comparison: Buprenorphine 1.0 mg TID vs Placebo; Test type: Other; p = 0.011, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 22.143, 95% CI 2-sided [5.46 to 38.83], Standard Error of Mean 8.1997

6. Secondary Outcome: NRS SPID Over 0 to 24 Hours After Time 0 (NRS SPID-24)
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug) and at multiple time points up to 24 hours after Time 0 (administration of first dose of study drug). Pain intensity difference is calculated by subtracting the pain intensity at each time point from the pain intensity at Time 0. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [maximum (max)=10 at each time point] and negative numbers indicate an increase in pain [minimum (min)=-10 at each time point]. The overall min and max are -10 and 10 times the number of hours specified; SPID-24 range is -240 to 240. The NRS SPID-24 was analyzed using an analysis of covariance (ANCOVA) model, which included treatment and site as main effects and Baseline pain intensity as the covariate.
Time Frame: Baseline and 0 to 24 hours after Time 0
Population: ITT Population included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 10
units on a scale | 83.668 (14.0612) | 70.071 (12.9115) | 76.666 (13.7558) | 19.787 (13.6231)
Statistical Analysis 1: Comparison: Buprenorphine 0.5 mg TID vs Placebo; Test type: Other; p = 0.001, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 63.881, 95% CI 2-sided [26.45 to 101.31], Standard Error of Mean 18.3971
Statistical Analysis 2: Comparison: Buprenorphine 1.0 mg BID vs Placebo; Test type: Other; p = 0.007, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 50.284, 95% CI 2-sided [14.48 to 86.09], Standard Error of Mean 17.5979
Statistical Analysis 3: Comparison: Buprenorphine 1.0 mg TID vs Placebo; Test type: Other; p = 0.004, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 56.879, 95% CI 2-sided [19.45 to 94.31], Standard Error of Mean 18.3984

7. Secondary Outcome: Percentage of Participants Who Used Rescue Medication for Pain
Description: The percentage of participants who needed to take an alternate medication for pain relief during the study.
Time Frame: From Time 0 (first dose of study drug) up to Day 9
Population: ITT Population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 10
percentage of participants | 44.4 | 54.5 | 60.0 | 100

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: from signing of informed consent to the Follow-up visit (up to 9 days). Non-serious Adverse Events: from the first dose of study drug to the Follow-up visit (up to 9 days).
Arm/Group | Buprenorphine 0.5 mg TID | Buprenorphine 1.0 mg BID | Buprenorphine 1.0 mg TID | Placebo
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/9 | 11/11 | 9/10 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buprenorphine 0.5 mg TID (N=9) | Buprenorphine 1.0 mg BID (N=11) | Buprenorphine 1.0 mg TID (N=10) | Placebo (N=10)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buprenorphine 0.5 mg TID (N=9) | Buprenorphine 1.0 mg BID (N=11) | Buprenorphine 1.0 mg TID (N=10) | Placebo (N=10)
Visual disturbance (Eye disorders) | 0 | 1 | 0 | 0
Burning mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Emesis (Gastrointestinal disorders) | 4 | 5 | 5 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Loose stools (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 10 | 7 | 3
Numbness mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Sore mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tingling lips (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tingling tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 3 | 0
Xerostomia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Shivering (General disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
Respiratory rate decreased (Investigations) | 0 | 0 | 1 | 0
Temperature elevation (Investigations) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Cramps in leg (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Low back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 4 | 4 | 0
Dizzy (Nervous system disorders) | 0 | 1 | 0 | 0
Drowsiness (Nervous system disorders) | 4 | 3 | 4 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 4 | 1 | 2
Intermittent headache (Nervous system disorders) | 0 | 0 | 0 | 2
Lightheadedness (Nervous system disorders) | 2 | 1 | 1 | 0
Paresthesia of fingers (Nervous system disorders) | 1 | 0 | 0 | 0
Shakiness (Nervous system disorders) | 0 | 0 | 1 | 0
Trembling (Nervous system disorders) | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Euphoria (Psychiatric disorders) | 0 | 1 | 0 | 0
Vivid dreams (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Singultus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Adhesive tape allergy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Diaphoresis (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Localised rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Pruritus facial (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Wheals (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early by the sponsor due to business reasons (40 participants enrolled out of 312 planned). Due to this early termination 10 outcome measures originally registered as pre-specified secondary are no longer secondaries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No